CLINICAL TRIAL: NCT00349531
Title: A Phase IV Randomised, Double-blind, Placebo-controlled, Dose Titration Trial With Pramipexole (Sifrol®, Mirapexin®) 0.125-0.75 mg/Day Per os for 12 Weeks to Investigate the Effects on RLS Symptoms (IRLS) and Sleep Disturbance (MOS Sleep Scale) in Out-patients With Idiopathic Restless Legs Syndrome
Brief Title: A Phase IV Trial With Pramipexole to Investigate the Effects on RLS Symptoms and Sleep Disturbance in Patients With RLS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Model: Parallel | Purpose: Treatment
Other Study IDs: 248.615
Record Dates: First submitted 2006-07-06; First posted 2006-07-07 (Estimated); Last update posted 2012-05-21 (Estimated); Status verified 2012-05

CONDITIONS: Restless Legs Syndrome
MeSH Terms: conditions — Restless Legs Syndrome | interventions — Pramipexole

INTERVENTIONS:
Drug: Pramipexole

SUMMARY:
The primary objective of this study is to investigate the effects on RLS symptoms and sleep disturbance of pramipexole (Mirapexin) 0.125 mg/day to 0.75 mg/day per os for 12 weeks, compared to placebo, in the treatment of patients with idiopathic Restless Legs Syndrome

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent consistent with ICH-GCP and local IRB/IEC requirements obtained prior to any study procedures being performed and the ability and willingness to comply with study treatment regimen and to attend study assessments.
2. Male or female out-patients aged 18-80 years.
3. Diagnosis of idiopathic RLS according to the clinical RLS criteria of the IRLSSG [P03-03355]. All four criteria must be present to fulfil the diagnosis of RLS:

   * An urge to move the legs, usually accompanied or caused by uncomfortable and unpleasant sensations in the legs. (Sometimes the urge to move is present without the uncomfortable sensations and sometimes the arms or other body parts are involved in addition to the legs)
   * The urge to move or unpleasant sensations begin or worsen during periods of rest or inactivity such as lying or sitting
   * The urge to move or unpleasant sensations are partially or totally relieved by movement, such as walking or stretching, at least as long as the activity continues
   * The urge to move or unpleasant sensations are worse in the evening or night than during the day or only occur in the evening or night. (When symptoms are very severe, the worsening at night may not be noticeable but must have been previously present).
4. RLS symptoms present at least 2 to 3 days per week during the last 3 months prior to baseline (Visit 2).
5. IRLS total score >15 at baseline (Visit 2).

Exclusion Criteria:

1. Women of child-bearing potential who do not use during the trial an adequate method of contraception.
2. Women of child-bearing potential not having negative pregnancy test at screening.
3. Breastfeeding women.
4. Concomitant or previous pharmacologic therapy for RLS with: dopamine agonists or levodopa (within 14 days prior to baseline), levodopa with augmentation, unsuccessful prior treatment with non-ergot dopamine agonists.
5. All treatment less than 14 days or concomitant treatment with medication or dietary supplements which could significantly influence RLS symptoms.
6. Withdrawal symptoms.
7. Pramipexole non-responders in other indications than RLS.
8. Patients with known hypersensitivity to pramipexole or any other component of the investigational product or placebo tablets.
9. Diabetes mellitus requiring insulin therapy.
10. Any of the following laboratory results at screening:

    * any clinically significant abnormalities in laboratory parameters;
    * haemoglobin below LLN.
11. Clinically significant renal disease or calculated creatinine clearance lower than 30 mL/minute.
12. Clinically significant hepatic disease or GPT >2 times the ULN.
13. Serum ferritin <10 ng/mL.
14. History of/or malignant melanoma.
15. History of/or clinically significant vision abnormalities.
16. History of/or any other sleep disorder (other than RLS-related).
17. History of/or major depressive disorder or any psychotic disorder, mental disorders or any present Axis I psychiatric disorder according to DSM IV requiring any medical therapy.
18. History of/or clinical signs of suicidal behaviour, suicide ideation or acute suicidal tendency according to the investigator's opinion.
19. History of/or alcohol abuse or drug addiction (within 2 years).
20. Patients on a shift-work-schedule or who are otherwise unable to follow a regular sleep-wake cycle.
21. Participation in an investigational drug study within one month.
22. Any clinically significant conditions that would interfere or constitute a health hazard for the patient.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 369 (Actual)
Dates: Start 2006-07; Primary Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Primary endpoint: change from baseline after 12 weeks in IRLS total score. Co-primary endpoint: change from baseline after 12 weeks in MOS sleep disturbance score. | 12 weeks after start of treatment

SECONDARY OUTCOMES:
Secondary endpoints: CGI-I and IRLS responder rate other MOS dimensions, RLS-6 items 4-6, IRLS item 10, VAS ,Verbal Fluency Tests ,RLS-QoL scores PGI responder rate adverse event profile, systolic and diastolic blood pressure, pulse rate | 12 weeks after start of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (49):
- Denmark (4):
  - 248.615.45103 Boehringer Ingelheim Investigational Site, Kongens Lyngby
  - 248.615.45102 Boehringer Ingelheim Investigational Site, København K
  - 248.615.45101 Boehringer Ingelheim Investigational Site, København NV
  - 248.615.45104 Boehringer Ingelheim Investigational Site, Vaerløse
- Finland (4):
  - 248.615.35101 Boehringer Ingelheim Investigational Site, Espoo
  - 248.615.35104 Boehringer Ingelheim Investigational Site, Joensuu
  - 248.615.35103 Boehringer Ingelheim Investigational Site, Lahti
  - 248.615.35102 Boehringer Ingelheim Investigational Site, Oulu
- Germany (9):
  - 248.615.49109 Boehringer Ingelheim Investigational Site, Berlin
  - 248.615.49105 Boehringer Ingelheim Investigational Site, Görlitz
  - 248.615.49108 Boehringer Ingelheim Investigational Site, Hattingen
  - 248.615.49106 Boehringer Ingelheim Investigational Site, München
  - 248.615.49102 Boehringer Ingelheim Investigational Site, Schwerin
  - 248.615.49103 Boehringer Ingelheim Investigational Site, Steglitz
  - 248.615.49101 Boehringer Ingelheim Investigational Site, Ulm
  - 248.615.49107 Boehringer Ingelheim Investigational Site, Witten
  - 248.615.49104 Boehringer Ingelheim Investigational Site, Würzburg
- Ireland (3):
  - 248.615.35302, Birr
  - 248.615.35301 Boehringer Ingelheim Investigational Site, Carrigtohill
  - 248.615.35303, Castlecomer
- Italy (8):
  - 248.615.39007 Policlinico di Bari - Università di Bari, Bari
  - 248.615.39006 Ospedale Civile di Dolo, Dolo (VE)
  - 248.615.39002 Ospedale S. Martino - A. O. Università di Genova, Genova
  - 248.615.39008 Policlinico Gaetano Martino, Messina
  - 248.615.39001 Istituto San Raffaele Turro, Milan
  - 248.615.39004 IRCCS Fondazione Istituto Neurologico "C. Mondino", Pavia
  - 248.615.39005 Ospedale S. Chiara, Pisa
  - 248.615.39003 A. O. Santa Maria della Misericordia, Udine
- Norway (5):
  - 248.615.47101 Boehringer Ingelheim Investigational Site, Bekkestua
  - 248.615.47102 Boehringer Ingelheim Investigational Site, Fevik
  - 248.615.47104 Boehringer Ingelheim Investigational Site, Moelv
  - 248.615.47103 Boehringer Ingelheim Investigational Site, Oslo
  - 248.615.47105 Boehringer Ingelheim Investigational Site, Tvedestrand
- Spain (6):
  - 248.615.3408 Hospital Nuestra Señora de Sonsoles, Ávila
  - 248.615.3402, Maderid
  - 248.615.3404 Hospital General Universitario Gregorio Marañón, Madrid
  - 248.615.3406, Madrid
  - 248.615.3407, Madrid
  - 248.615.3403 Hospital General de Catalunya, San Cugat Del Valles (Barcelona)
- Sweden (4):
  - 248.615.46101 Boehringer Ingelheim Investigational Site, Gothenburg
  - 248.615.46103 Boehringer Ingelheim Investigational Site, Gothenburg
  - 248.615.46102 Boehringer Ingelheim Investigational Site, Hedemora
  - 248.615.46104 Boehringer Ingelheim Investigational Site, Örebro
- United Kingdom (6):
  - 248.615.44006 Boehringer Ingelheim Investigational Site, Buckshaw Village, Chorley
  - 248.615.44004 Boehringer Ingelheim Investigational Site, Cambridge
  - 248.615.44007 Boehringer Ingelheim Investigational Site, Manchester
  - 248.615.44009 Boehringer Ingelheim Investigational Site, Reading
  - 248.615.44002 Boehringer Ingelheim Investigational Site, Romford
  - 248.615.44005 Boehringer Ingelheim Investigational Site, West Green, Crawley

REFERENCES:
- [Derived] Hornyak M, Sohr M, Busse M; 604 and 615 Study Groups. Evaluation of painful sensory symptoms in restless legs syndrome: experience from two clinical trials. Sleep Med. 2011 Feb;12(2):186-9. doi: 10.1016/j.sleep.2010.11.007. Epub 2011 Jan 21. PMID 21256799